CLINICAL TRIAL: NCT01366807
Title: Screening of Nutritional Status and Predictors of Adverse Outcome in Cardiac Surgery
Brief Title: Screening of Nutritional Status in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Efremov Sergey, Anesthesist, Meshalkin Research Institute of Pathology of Circulation
Other Study IDs: SCR2011
Record Dates: First submitted 2011-05-31; First posted 2011-06-06 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, white cells
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Screening of nutritional status is unsolved problem in cardiac surgery. Applicability of such criteria as body mass index and albumin and screening scales (MNA, NRS-2002, SGA, SNAQ) in cardiac surgery is controversial and insufficiently studied. Furthermore, there is some known predictors of poor outcome, which closely related to nutritional status (C-reactive protein, total lymphocyte count). The aim of this study is assessment of several nutritional screening scales, objective nutritional criteria and predictors for the purpose of detection of most informative one or its combination.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with cardiovascular disease operated on under cardiopulmonary bypass

Exclusion Criteria:

* Age under 18 years
* Emergency
* Participation in other trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, who live in Russia, mostly in Siberia whom scheduled to cardiac surgery in one institution.
Sampling Method: Probability Sample
Enrollment: 1210 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Mortality | Participants will be followed for the duration of hospital stay, an average of 4 weeks.

SECONDARY OUTCOMES:
Complications | Participants will be followed for the duration of hospital stay, an average of 4 weeks.
  Postoperative cardiac failure, infectious complications, clinically significant arrhythmia, bleeding
Intensive care unit stay | Participants will be followed for the duration of hospital stay, an average of 4 weeks.
Hospital stay | Participants will be followed for the duration of hospital stay, an average of 4 weeks.
Ventilation time | Participants will be followed for the duration of hospital stay, an average of 4 weeks.
  Period between admission to ICU after the surgery and extubation

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir V Lomivorotov, MD, PhD, Principal Investigator — Novosibirsk Research Institute of Pathology of Circulation
Locations (1):
- Novosibirsk Research Institute of Patholgy of Circulation, Novosibirsk, Russia

REFERENCES:
- [Background] Lomivorotov VV, Efremov SM, Boboshko VA, Leyderman IN, Lomivorotov VN, Cheung AT, Karaskov AM. Preoperative total lymphocyte count in peripheral blood as a predictor of poor outcome in adult cardiac surgery. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):975-80. doi: 10.1053/j.jvca.2010.12.006. Epub 2011 Feb 26. PMID 21354824
- [Result] Lomivorotov VV, Efremov SM, Boboshko VA, Nikolaev DA, Vedernikov PE, Lomivorotov VN, Karaskov AM. Evaluation of nutritional screening tools for patients scheduled for cardiac surgery. Nutrition. 2013 Feb;29(2):436-42. doi: 10.1016/j.nut.2012.08.006. Epub 2012 Nov 27. PMID 23200301